CLINICAL TRIAL: NCT01439009
Title: A Multi-center,_double-blind,_pararel-group Comparison Trial to Investigate the Effect of Short-term Administration of Tolvaptan on Mid- to Long-term Prognosis of Heart Failure Patients (Phase_4 Study)
Brief Title: Effect of Tolvaptan on Mid- to Long-term Prognosis of Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-10-005; JapicCTI-111621 (Other: JAPIC)
Record Dates: First submitted 2011-09-15; First posted 2011-09-22 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Volume overload; Tolvaptan; loop diuretics
MeSH Terms: conditions — Heart Failure; Edema | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental): 15 mg
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo of tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Once-daily oral administration of one tolvaptan 15 mg tablet in the morning
  Arms: Tolvaptan
Drug: Placebo of tolvaptan — Once-daily oral administration of one placebo tablet in the morning
  Arms: Placebo

SUMMARY:
One tolvaptan 15 mg tablet or placebo tablet will be orally administered once daily in the morning for up to 14 days to heart failure patients with volume overload that does not show adequate response to other diuretics such as loop diuretics in order to investigate the effect of tolvaptan on the mid- to long-term prognosis of the target population. The efficacy of tolvaptan during the treatment period will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients from whom informed consent has been properly obtained in writing prior to start of the trial
* Patients who have been clinically diagnosed with heart failure
* Patients with any of the following conditions or symptoms: lower limb edema, dyspnea, jugular venous distension, hepatomegaly, pulmonary rales, third heart sound, or pulmonary congestion
* Patients who have been receiving loop diuretics, thiazide diuretics, or anti-aldosterone diuretics
* Male or female patients of age 20 to 85 years inclusive (at time of informed consent)
* Patients who, together with their partner(s), are able to use an appropriate method of contraception until 3 months after final trial drug administration
* Patients who are able to be hospitalized at the trial site for at least 7 days from the start of trial drug administration

Exclusion Criteria:

* Patients with a history of hypersensitivity to any ingredient of the drug or to tolvaptan analogues (e.g., mozavaptan hydrochloride)
* Patients with anuria
* Patients who cannot sense thirst or who have difficulty with fluid intake
* Patients with hypernatremia (serum sodium concentration > institutional upper limit of normal) 5) Female patients who are pregnant, possibly pregnant, or nursing
* Patients judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial due to any of the following conditions or symptoms:

  * Hyponatremia (serum sodium concentration < 125 mEq/L)
  * Serious coronary artery disease or cerebrovascular disease
  * Hyperkalemia
  * Severe renal disorder
  * Poorly controlled diabetes mellitus
  * Severe hepatic disease
  * Impaired urinary excretion due to urinary stenosis, calculus, or tumor
  * Cardiac valve disease with significant heart valve stenosis
  * Malignant tumor of unfavorable prognosis
* Patients with suspected hypovolemia
* Patients with an implanted circulatory support device
* Patients in whom acute cardiac infarction occurred within 30 days prior to the screening examination
* Patients who participated in any other clinical trial or postmarketing clinical trial within 30 days prior to the date of informed consent for the present trial
* Patients who received tolvaptan within 26 weeks prior to the date of informed consent
* Patients who are otherwise judged by the investigator or sub-investigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chube Region
  - Chushikoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tolvaptan | Placebo
Started | 50 | 50
Completed | 42 | 47
Not Completed | 8 | 3
Not completed — Physician Decision | 5 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Deviation of exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 22
  >=65 years | 41 | 37 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (8.4) | 71.7 (11.2) | 72.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 29 | 37 | 66
Region of Enrollment [Number; unit: participants]
  Japan | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Cummulative Incidence of Events at Week 26
Description: From start day of IMP administration to final day of follow up period, 1) and 2) below were defined as event
  1. Death from cardiovascular events
  2. Worsening of heart failure
     * The day of re-hospitalization due to worsening of heart failure
     * The day of medication below due to worsening of heart failure Phosphodiesterase III inhibitors (Injection), Catecholamine preparations (Injection), Colforsin preparations (Injection), Diuretics (Injection), Human atrial natriuretic peptide preparations (Injection)：Calperitide (Injection)
Time Frame: Week 26
Measure: Number; unit: Percentage of events at 26 weeks
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 50 | 50
Percentage of events at 26 weeks | 35.6 | 43.8

2. Primary Outcome: Mortality （Number of Death）
Description: Statistical comparison was not done.
Time Frame: Week26
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 50 | 50
participants | 2 | 3

3. Primary Outcome: Body Weight
Description: The comparison of the average of amount of change from baseline. Statistical comparison was not done.
Time Frame: Day15
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 47 | 44
kg | -1.99 (1.61) | -1.20 (1.97)

4. Primary Outcome: Number of Subjects Whose Lower Limb Edema Severity Grading Improved by One or More Grade
Description: Of the subjects who had lower limb edema at baseline, the number of subjects whose lower limb edema severity grading. Statistical comparison was not done.
Time Frame: Day15
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 35 | 25
participants | 27 | 16

5. Primary Outcome: Jugular Venous Distension
Description: The comparison of the average of amount of change from baseline. Statistical comparison was not done.
Time Frame: Day15
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 47 | 43
cm | -0.94 (2.07) | -1.23 (2.78)

6. Primary Outcome: Change in Liver Size From Baseline
Description: The comparison of the average of amount of change from baseline. Statistical comparison was not done．
Time Frame: Day15
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 47 | 43
cm | -0.20 (0.52) | -0.19 (0.55)

7. Primary Outcome: Pulmonary Rales
Description: Of the subjects who had pulmonary rales at baseline, the number of subjects whose symptom was resolved at completion of treatment. Statistical comparison was not done.
Time Frame: Day15
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 16 | 17
participants | 13 | 9

8. Primary Outcome: Third Heart Sound
Description: Of the subjects who had third heart sound at baseline, the number of subjects whose symptom was resolved at completion of treatment. Statistical comparison was not done.
Time Frame: Day15
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 14 | 16
participants | 8 | 10

9. Primary Outcome: Cardiothoracic Ratio
Description: Investigator majored Thoracic length and Cardiac length from chest X-ray. Cardiothoracic Ratio was calculated from Cardiac length/Thoracic length*100. Lowering of Cardiothoracic Ratio suggests recovery from heart congestion.
  The comparison of the average of amount of change from baseline. Statistical comparison was not done.
Time Frame: Day15
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 47 | 44
Percentage | -2.13 (3.53) | -0.83 (3.85)

10. Primary Outcome: Pulmonary Congestion
Description: Of the subjects who had pulmonary congestion at baseline, the number of subjects whose pulmonary congestion severity grading showed an improvement of one grade or more (eg, moderate to mild) at completion of treatment. Statistical comparison was not done.
Time Frame: Day15
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 40 | 42
participants | 24 | 20

11. Primary Outcome: Plasma Brain Natriuretic Peptide (BNP) Concentration
Description: The comparison of the average of amount of change from baseline. Statistical comparison was not done.
Time Frame: Day15
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 46 | 44
pg/mL | -72.60 (268.90) | -166.96 (353.34)

12. Primary Outcome: Dypnea
Description: Of the subjects who had dyspnoea at baseline, the number of subjects whose symptom was resolved at completion of treatment. Statistical comparison was not done.
Time Frame: Day15
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 15 | 20
participants | 11 | 12

13. Primary Outcome: Number of Subjects Whose New York Heart Association (NYHA) Classification Improved by One More Grade From Baseline
Description: New York Heart Association (NYHA) Classification is below ClassI：No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  ClassII：Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  ClassIII：Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  ClassIV：Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: The day after last IMP administration and Baseline
Measure: Number; unit: participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 47 | 44
participants | 22 | 24

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Tolvaptan | Placebo
Serious Adverse Events (participants affected / at risk) | 24/50 | 22/50
Other Adverse Events (participants affected / at risk) | 31/50 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=50) | Placebo (N=50)
Cardiac failure (Cardiac disorders) | 13 | 19
Acute Cardiac Failure (Cardiac disorders) | 0 | 1
Congestive Cardiac Failure (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diabetic retina edema (Eye disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Rhinopharyngitis (Infections and infestations) | 0 | 1
Pneumoria (Infections and infestations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=50) | Placebo (N=50)
Constipation (Gastrointestinal disorders) | 6 | 2
Thirst (General disorders) | 10 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Blood potassium increased (Investigations) | 3 | 1
Blood sodium increased (Investigations) | 8 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No